CLINICAL TRIAL: NCT05189522
Title: Innova Breeze®-Based Roadmap for Peripheral Arterial Disease
Acronym: IBREED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBREED
Record Dates: First submitted 2021-12-29; First posted 2022-01-12 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Innova Breeze®-based roadmap (Experimental): An Innova Breeze® bolus chase acquisition is realized prior to the revascularization to assess the lesions of the entire target limb. Guidance to the different lesions is done using a 2D roadmap based on the Innova Breeze® bolus acquisition frames if the patient position has not moved on the table.
  An Innova Breeze® bolus chase acquisition is realized to assess the final result of the revascularization of the target limb. Both Innova Breeze® bolus chases are required at field of view 30-cm. Finally, the sheath is retrieved and the hemostasis at the puncture site is realized via a manual compression or using a vascular closure device.
  DSAs are performed with the injector set at 7mL/s and the volume at 7mL (pressure limit 1000psi) for femoropopliteal assessment. Innova Breeze® bolus chase acquisitions are performed with the injector set at 4mL/s and the volume at 24mL (pressure limit 1000psi). An injector with iodinated contrast (50% of dilution) will be used.
  Interventions: Device: Innova Breeze®-based roadmap
- control group (Other): 2D roadmap guidance is used based on DSA. The treatment of the target lesion is let at the physician discretion. Treatment result of each lesion is checked by a DSA with 1 incidence.
  After treatment overall limb assessment will be done through multiple staged DSA.
  Finally, the sheath is retrieved and the hemostasis at the puncture site is realized via a manual compression or using a vascular closure device.
  DSAs are performed with the injector set at 7mL/s and the volume at 7mL (pressure limit 1000psi) for femoropopliteal assessment. An injector with iodinated contrast (50% of dilution) will be used.
  For hospitalized patients, three to five days after the procedure, a blood test is performed to assess the eGFR, as part of the usual care of patients. If the patient is no longer hospitalized, at the time of this examination, the investigating physician has given him an order before his discharge to perform this examination in an analysis laboratory.
  Interventions: Other: Control Group

INTERVENTIONS:
Device: Innova Breeze®-based roadmap — An Innova Breeze® bolus chase acquisition is realized to assess the final result of the Revascularization of the target limb. Both Innova Breeze® bolus chases are required at field of view 30-cm
  Arms: Innova Breeze®-based roadmap
Other: Control Group — 2D roadmap guidance is used based on DSA. The treatment of the target lesion is let at the physician discretion. Treatment result of each lesion is checked by a DSA with 1 incidence.
  After treatment overall limb assessment will be done through multiple staged DSA.
  Finally, the sheath is retrieved and the hemostasis at the puncture site is realized via a manual compression or using a vascular closure device.
  DSAs are performed with the injector set at 7mL/s and the volume at 7mL (pressure limit 1000psi) for femoropopliteal assessment. An injector with iodinated contrast (50% of dilution) will be used.
  For hospitalized patients, three to five days after the procedure, a blood test is performed to assess the eGFR, as part of the usual care of patients. If the patient is no longer hospitalized, at the time of this examination, the investigating physician has given him an order before his discharge to perform this examination in an analysis laboratory.
  Arms: control group

SUMMARY:
Over the past decade, interventional endovascular treatment, whenever feasible, has become the first line management in the treatment of lower extremity arterial disease (LEAD) for many indications. Growth of endovascular therapy was based on shorter hospital length of stay and lower complications rates. This minimally invasive procedure allows the revascularization of the lower limbs under fluoroscopy guidance, with injection of iodinated contrast allowing to analyze the arteries. However, many of these patients present renal insufficiency which could be worsened due to the iodinated contrast injections during the endovascular procedure for LEAD. Consequently, the vascular interventionalist should find a way to achieve patient revascularization while minimizing iodinated contrast injections in order to maintain the renal function.

The aim of this study is to compare the amount of iodine contrast used during LEAD endovascular revascularization with and without the Innova Breeze® and blended roadmap software.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years
* Patient has a history of symptomatic peripheral arterial disease (Rutherford classification 2-6)
* Patients with indication of femoropopliteal revascularization according the European guidelines (1)
* Patient agrees to undergo all protocol required follow-up examinations and requirements at the investigational site
* French-speaking patient
* Patient is affiliated to the Social Security or equivalent system
* Patients is able and willing to give free, informed and express oral consent
* Iliac and/or below the knee lesions are allowed in combination to femoropopliteal lesions

Exclusion Criteria:

* Upper limb approach
* Femoral antegrade approach
* Pregnant or breastfeeding woman
* Adult under guardianship or trusteeship
* Iodinated contrast allergy
* Reduction in estimated Glomerular Filtration Ratio (eGFR) ≤ 29 ml/min/m2 (11)
* Patients included in other studies which interact with intraoperative imaging protocols
* Concurrent participation in an interventional (drug or device) study for which the follow-up period is not complete.
* Patient under tutorship or curatorship
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2024-02-10 (Estimated); Study Completion 2024-05-25 (Estimated)

PRIMARY OUTCOMES:
Amount of iodinated contrast volume | Day 1
  This outcome corresponds to the volume of iodinated contrast used at the end of the procedure.

SECONDARY OUTCOMES:
Patient safety in terms of radiation exposure at the end of the procedure | Day 1
  This outcome corresponds to the number of DSA runs.
Staff safety in terms of radiation exposure at the end of the procedure | Day 1
  This outcome corresponds to the Operator exposure (Sv).
Patient clinical improvement | Month 1
  This outcome corresponds to the clinical status (Rutherford stage).
Estimation of renal function post-operative | Day 4
  This outcome corresponds to the Glomerular filtration rate (GFR).
Estimation of renal function at 1 month | Month 1
  This outcome corresponds to the Glomerular filtration rate (GFR)

CONTACTS AND LOCATIONS:
Overall Officials: Yann GOUEFFIC, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, Collet JP, Czerny M, De Carlo M, Debus S, Espinola-Klein C, Kahan T, Kownator S, Mazzolai L, Naylor AR, Roffi M, Rother J, Sprynger M, Tendera M, Tepe G, Venermo M, Vlachopoulos C, Desormais I; ESC Scientific Document Group. 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS): Document covering atherosclerotic disease of extracranial carotid and vertebral, mesenteric, renal, upper and lower extremity arteriesEndorsed by: the European Stroke Organization (ESO)The Task Force for the Diagnosis and Treatment of Peripheral Arterial Diseases of the European Society of Cardiology (ESC) and of the European Society for Vascular Surgery (ESVS). Eur Heart J. 2018 Mar 1;39(9):763-816. doi: 10.1093/eurheartj/ehx095. No abstract available. PMID 28886620
- [Background] Fowkes FG, Rudan D, Rudan I, Aboyans V, Denenberg JO, McDermott MM, Norman PE, Sampson UK, Williams LJ, Mensah GA, Criqui MH. Comparison of global estimates of prevalence and risk factors for peripheral artery disease in 2000 and 2010: a systematic review and analysis. Lancet. 2013 Oct 19;382(9901):1329-40. doi: 10.1016/S0140-6736(13)61249-0. Epub 2013 Aug 1. PMID 23915883
- [Background] Criqui MH, Matsushita K, Aboyans V, Hess CN, Hicks CW, Kwan TW, McDermott MM, Misra S, Ujueta F; American Heart Association Council on Epidemiology and Prevention; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Radiology and Intervention; Council on Lifestyle and Cardiometabolic Health; Council on Peripheral Vascular Disease; and Stroke Council. Lower Extremity Peripheral Artery Disease: Contemporary Epidemiology, Management Gaps, and Future Directions: A Scientific Statement From the American Heart Association. Circulation. 2021 Aug 31;144(9):e171-e191. doi: 10.1161/CIR.0000000000001005. Epub 2021 Jul 28. PMID 34315230
- [Background] Criqui MH, Aboyans V. Epidemiology of peripheral artery disease. Circ Res. 2015 Apr 24;116(9):1509-26. doi: 10.1161/CIRCRESAHA.116.303849. PMID 25908725
- [Background] O'Hare AM, Glidden DV, Fox CS, Hsu CY. High prevalence of peripheral arterial disease in persons with renal insufficiency: results from the National Health and Nutrition Examination Survey 1999-2000. Circulation. 2004 Jan 27;109(3):320-3. doi: 10.1161/01.CIR.0000114519.75433.DD. Epub 2004 Jan 19. PMID 14732743
- [Background] Ungprasert P, Pornratanarangsi S. Correlation between peripheral arterial disease and stage of chronic kidney disease. J Med Assoc Thai. 2011 Feb;94 Suppl 1:S46-50. PMID 21728271
- [Background] Amighi J, Schlager O, Haumer M, Dick P, Mlekusch W, Loewe C, Bohmig G, Koppensteiner R, Minar E, Schillinger M. Renal artery stenosis predicts adverse cardiovascular and renal outcome in patients with peripheral artery disease. Eur J Clin Invest. 2009 Sep;39(9):784-92. doi: 10.1111/j.1365-2362.2009.02180.x. Epub 2009 Jun 12. PMID 19522837
- [Background] Andreucci M, Faga T, Serra R, De Sarro G, Michael A. Update on the renal toxicity of iodinated contrast drugs used in clinical medicine. Drug Healthc Patient Saf. 2017 May 22;9:25-37. doi: 10.2147/DHPS.S122207. eCollection 2017. PMID 28579836